CLINICAL TRIAL: NCT00712348
Title: A Phase 3 Multicenter, Open-label, Switchover Trial to Assess the Safety and Efficacy of Plant Cell Expressed Recombinant Human Glucocerebrosidase in Patients With Gaucher Disease Treated With Imiglucerase
Brief Title: Switchover Trial From Imiglucerase to Plant Cell Expressed Recombinant Human Glucocerebrosidase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-06-002
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Gaucher Disease
Keywords: Gaucher disease; imiglucerase; glucocerebrosidase; enzyme replacement therapy; lysosomal storage disorder
MeSH Terms: conditions — Gaucher Disease; Lysosomal Storage Diseases | interventions — taliglucerase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Taliglucerase alfa (Experimental): Open label taliglucerase alfa treatment
  Interventions: Drug: Taliglucerase alfa

INTERVENTIONS:
Drug: Taliglucerase alfa — Intravenous infusion every 2 weeks
  Other Names: Plant cell expressed recombinant glucocerebrosidase (prGCD)

SUMMARY:
This is a multi-center, open-label, switchover trial to assess the safety of taliglucerase alfa in 30 patients with Gaucher disease who are currently being treated with imiglucerase (Cerezyme®) enzyme replacement therapy.

DETAILED DESCRIPTION:
This is a multi-center, open-label, switchover trial to assess the safety of taliglucerase alfa in 30 patients with Gaucher disease who are currently being treated with imiglucerase (Cerezyme®) ERT. Eligible patients will enter a 12-week Stability Evaluation Period to establish the stability of their disease. Patients with stable disease will then be switched from their imiglucerase treatment to receive intravenous (IV) infusions of taliglucerase alfa every two weeks for a total of 20 IV infusions. The dose of taliglucerase alfa will be equal to each patient's previous imiglucerase dose. The infusions will be administered at the selected investigational site (clinic/hospital), infusion center, or at home. At the end of the 9-month treatment period (20 visits, 38 weeks) eligible patients will be offered enrollment in an open-label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 2 years or older
* Confirmed diagnosis of Gaucher disease by the enzymatic activity assay
* Stable Gaucher disease
* Treatment with imiglucerase (Cerezyme®) for at least 2 years and on a stable maintenance regimen (dose and regimen unchanged, except for situation of drug shortage) for at least the last six months
* Able to provide written informed consent

Exclusion Criteria:

* Currently taking another experimental drug for any condition
* History of allergy to carrots
* History of allergy to beta lactam antibiotics
* Previous infusion reaction suspected to be allergic in nature to Cerezyme® or Ceredase® or receiving premedication to prevent infusion reactions
* Presence of HIV and/or HBsAg and/or hepatitis C infection
* Presence of unresolved anemia due to iron, folic acid or vitamin B12 deficiency
* Presence of any significant comorbidity that could confound the interpretation of the clinical response to taliglucerase alfa
* Presence of any medical, emotional, behavioral or psychological condition that in the judgment of the Investigator would interfere with the patient's compliance with the requirements of the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-12; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (3):
  - University Research Foundation for Lysosomal Storage Diseases, Inc., Coral Springs, Florida
  - Department of Human Genetics, Emory University School of Medicine, Decatur, Georgia
  - Neurogenetics, NYU at Rivergate, New York, New York
- Bone Marrow Transplant Service, The Royal Melbourne Hospital, Parkville, Victoria, Australia
- Mount Sinai Hospital, Toronto, Ontario, Canada
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
- Sala de Hematologia, Hospital Universitario Miguel Servet, Zaragoza, Spain
- United Kingdom (2):
  - Lysosomal Disorders Service, Addenbrookes Hospital NHS Trust, Cambridge
  - Royal Free Hospital, London

REFERENCES:
- [Derived] Pastores GM, Petakov M, Giraldo P, Rosenbaum H, Szer J, Deegan PB, Amato DJ, Mengel E, Tan ES, Chertkoff R, Brill-Almon E, Zimran A. A Phase 3, multicenter, open-label, switchover trial to assess the safety and efficacy of taliglucerase alfa, a plant cell-expressed recombinant human glucocerebrosidase, in adult and pediatric patients with Gaucher disease previously treated with imiglucerase. Blood Cells Mol Dis. 2014 Dec;53(4):253-60. doi: 10.1016/j.bcmd.2014.05.004. Epub 2014 Jun 18. PMID 24950666

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Taliglucerase Alfa
Started | 31
Completed | 30
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 25
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
  Canada | 1
  Spain | 4
  Australia | 3
  Israel | 9
  United Kingdom | 2
  Serbia | 4
  Singapore | 1
Religion [Number; unit: participants]
  JEWISH - ASHKENAZI | 14
  JEWISH - NONASHKENAZI | 0
  NON JEWISH | 15
  UNREPORTED | 2

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Platelet Count
Time Frame: Every 3 months from Baseline to Month 9
Measure: Mean (Standard Deviation); unit: platelets/mm^3
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 30
platelets/mm^3
  Baseline | 161137 (73387)
  Month 3 | 150800 (66038)
  Month 6 | 157586 (78357)
  Month 9 | 161167 (80820)

2. Other Pre Specified Outcome: Spleen Volume
Description: Spleen volume measured by MRI in mL
Time Frame: Baseline and 9 Months
Population: 25 patients had spleen volume measured by MRI, 2 were MRI phobic and 3 were splenectomized
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 25
mL
  Baseline | 720.5 (579.5)
  Month 9 | 654.7 (535.9)

3. Other Pre Specified Outcome: Liver Volume
Description: Liver volume measured by MRI
Time Frame: Baseline and 9 months
Population: 2 patients were MRI phobic
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 28
mL
  Baseline | 1766 (474.5)
  Month 9 | 1716 (455.6)

4. Primary Outcome: Hemoglobin
Time Frame: Every 3 months from Baseline to Month 9
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Taliglucerase Alfa
Number analyzed (Participants) | 30
g/dL
  Baseline | 13.5 (1.4)
  Month 3 | 13.3 (1.5)
  Month 6 | 13.3 (1.6)
  Month 9 | 13.4 (1.5)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Taliglucerase Alfa
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taliglucerase Alfa (N=31)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Right nostril due to perforated septum - Not Related
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) — Not Related
PELVIC PROLAPSE (Reproductive system and breast disorders) | 1 (1) — Prolapsed rectum, cervix and bladder - Not Related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taliglucerase Alfa (N=31)
DIARRHOEA (Gastrointestinal disorders) | 2 (2)
PAIN (General disorders) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3)
HEADACHE (Nervous system disorders) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No